CLINICAL TRIAL: NCT04055597
Title: Effects of Upper Extremity Rehabilitation Robot and Transcranial Direct Current Stimulation on Upper Extremity Function Among Subjects With Tremor After Cerebellar and Brainstem Stroke
Brief Title: Effects of Upper Extremity Rehabilitation Robot and Transcranial Direct Current Stimulation Among Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRC-2017-01-004
Record Dates: First submitted 2018-03-01; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Stroke
Keywords: cerebellar stroke; upper extremity rehabilitation robot; transcranial direct current stimulation; stroke rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot and tDCS on-line (Experimental): Combined transcranial direct current stimulation(tDCS) on-line and upper extremity rehabilitation robot
  Interventions: Other: Robot and tDCS on-line
- Robot and sham tDCS (Sham Comparator): Combined sham tDCS and upper extremity rehabilitation robot
  Interventions: Other: Robot and sham tDCS

INTERVENTIONS:
Other: Robot and tDCS on-line — Combined transcranial direct current stimulation(tDCS) on-line and upper extremity rehabilitation robot for 5 times a week for 4 weeks
  Arms: Robot and tDCS on-line
Other: Robot and sham tDCS — Combined sham tDCS and upper extremity rehabilitation robot for 5 times a week for 4 weeks
  Arms: Robot and sham tDCS

SUMMARY:
Effects of upper extremity rehabilitation robot and transcranial direct current stimulation on upper extremity function among subjects with tremor after stroke

ELIGIBILITY:
Inclusion Criteria:

* Stroke with cerebellar hemorrhage or infarction
* ataxia or tremor on upper extremities secondary to stroke
* Cognitively intact enough to understand and follow the instructions from the investigator

Exclusion Criteria:

* History of surgery of affected upper limb
* Fracture of affected upper limb

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Scale for the assessment and rating of ataxia | Change of Scale for the assessment and rating of ataxia at 4 weeks after baseline compared to baseline
  Change of Scale for the assessment and rating of ataxia
Change of Functional ataxia rating scale - upper limb | Change of the Functional ataxia rating scale - upper limb, at 4 weeks after baseline compared to baseline
  Change of Functional ataxia rating scale - upper limb

SECONDARY OUTCOMES:
Fugl-Meyer Assessment - upper extremity | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Fugl-Meyer Assessment - upper extremity
Composite cerebellar functional severity score | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Composite cerebellar functional severity score (Nine hole peg test + click test)
Jerk during reaching and finger pointing | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Kinematic data during reaching and finger pointing using Trakstar
Smoothness during reaching and finger pointing | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Kinematic data during reaching and finger pointing using Trakstar
Behavioral activation system/behavioral inhibition system scale | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  In terms of motivation
Beck's depression index | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Beck's depression index
Stroke rehabilitation motivation scale | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Stroke rehabilitation motivation scale
Intrinsic motivation inventory | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Intrinsic motivation inventory
Numeric rating scale for upper extremity pain | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Question about the upper extremity pain (0-10; higher is better)
Functional reaching test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Functional reaching test
modified Barthel index | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  modified Barthel index
% maximal voluntary contraction from upper extremity muscles during reaching task | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  data from surface electromyography from upper extremity muscles during reaching task
Kinematic data during scale for the assessment and rating of ataxia | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Kinematic data during scale for the assessment and rating of ataxia
Scale for the assessment and rating of ataxia | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Scale for the assessment and rating of ataxia
Functional ataxia rating scale - upper limb | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Functional ataxia rating scale - upper limb, kinematic data during scale for the assessment
Kinematic data during scale during the Functional ataxia rating scale - upper limb | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Kinematic data during scale during the Functional ataxia rating scale - upper limb

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, South Korea